CLINICAL TRIAL: NCT00941759
Title: A Prospective Analysis of Surgery in Patients Presenting With Stage IV Breast Cancer
Brief Title: Analysis of Surgery in Patients Presenting With Stage IV Breast Cancer
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: University of Chicago (Other); Dana-Farber Cancer Institute (Other); Georgetown University (Other); Johns Hopkins University (Other); M.D. Anderson Cancer Center (Other); University of Alabama at Birmingham (Other); University of California, San Francisco (Other); University of North Carolina (Other); Duke University (Other); Vanderbilt-Ingram Cancer Center (Other); Indiana University Melvin and Bren Simon Cancer Center (Other); Mayo Clinic (Other); University of Pittsburgh Medical Center (Other); University of Michigan (Other)
Responsible Party: Sponsor
Other Study IDs: 09-056
Record Dates: First submitted 2009-07-16; First posted 2009-07-20 (Estimated); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
Keywords: Breast; Blood and tissue collection; Epidemiologic; Questionnaire; TBCRC (Translational Breast Cancer Research Consortium); 09-056
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and tissue collection

GROUPS / COHORTS (2):
- Known or suspected Stage IV disease & an intact primary: Pt will be asked to undergo a research core needle biopsy of the primary tumor. If pts are not agreeable to a research biopsy then the original diagnostic biopsy material will be requested. They will also undergo a diagnostic biopsy of a metastatic site, if not already performed, and a blood draw as appropriate for correlative science studies. Additionally, patients will complete a general medical questions form at the time of enrollment.
- Unsuspected metastatic disease W/I 3 months of primary b: A blood sample will be collected and patients will complete a general medical questions form at the time of enrollment. Paraffin tissue from the prior surgical procedure will be obtained as Tissue sample. Paraffin tissue from the diagnostic biopsy of a metastatic site will also be obtained. In the event that fresh frozen tissue is available for either site this will also be requested.

SUMMARY:
The purpose of this study is to study patients presenting with stage IV breast cancer. Stage IV means that the breast cancer has spread to another part of the body outside the breast. This study is important because in different parts of the country some patients are being offered surgical treatment for the breast tumor and some are not. The doctors do not know if surgery for the breast tumor is helpful in patients with stage IV breast cancer. The doctors will collect information about the patient and their treatment to learn more about how patients and doctors make treatment decisions. The doctor will also collect blood samples and tissue samples for laboratory studies to learn more about tumors that have spread to other parts of the body.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Known or suspected Stage IV breast cancer with intact primary tumor
* Known or suspected Stage IV breast cancer with intact primary tumor, having begun systemic therapy within the past 12 months
* Known or suspected Stage IV breast cancer within 3 months of local breast surgery
* Known or suspected Stage IV breast cancer within 3 months of local breast surgery, having begun systemic therapy within the past 12 months

Exclusion Criteria:

* Primary breast cancer diagnosis made by FNA only and no pre-treatment core biopsy planned for diagnostic or research purposes.
* Failure of MSKCC or participating site to confirm Stage IV breast cancer diagnosis by biopsy within 30 days of study enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential research subjects will be identified by a member of the patient's treatment team, either at the time of consultation with the breast surgeon or breast medical oncologist. Patients will be accrued from each of the 15 participating sites.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-07; Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
Measure response to first-line therapy, frequency of surgical referral and the proportion of patients who undergo surgery of the primary tumor in stage IV disease. | 2 years

SECONDARY OUTCOMES:
Determine the incidence of uncontrolled local disease in patients who do/do not undergo surgery. | 2 years
Correlate molecular characteristics of the primary tumor with conventional prognostic factors and survival in patients presenting with stage IV breast cancer. | 2 years
Perform correlative molecular studies of circulating tumor cells, primary and metastatic tumor samples in stage IV breast cancer. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Monica Morrow, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (20):
- United States (20):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California San Francisco, San Francisco, California
  - Georgetown University, Washington D.C., District of Columbia
  - Washington Cancer Institute at Washington, Washington D.C., District of Columbia
  - University of Chicago, Chicago, Illinois
  - The Indiana University Simon Cancer Center, Indianapolis, Indiana
  - John Hopkins Medical Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - University of North Carolina School of Medicine, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Md Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org